CLINICAL TRIAL: NCT03599141
Title: Pilot RCT to Evaluate the Effects of a Trust-Building Depression Management Intervention on Moderate Depressive Symptoms in Low-Income Adolescents
Brief Title: Testing TRUST Depression Management Intervention
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Heather K. Hardin, PhD, RN, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180519; U54MD002265-11 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-07-26 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms; Quality of Life
Keywords: adolescent; parent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depression Management (Active Comparator): 8 weekly group sessions
  Interventions: Behavioral: Depression Management
- Trust-building Self-management Together (Experimental): 8 weekly group sessions
  Interventions: Behavioral: Trust-building Self-management Together

INTERVENTIONS:
Behavioral: Trust-building Self-management Together — Trust building plus depression self-management
  Arms: Trust-building Self-management Together
Behavioral: Depression Management — Traditional depression self-management
  Arms: Depression Management

SUMMARY:
This study evaluates the effectiveness of a novel depression self-management intervention in adolescents with depression.

DETAILED DESCRIPTION:
Half of participants will receive a traditional depression self-management intervention, while the other half will receive the novel depression self-management intervention. In an exploratory, pilot 2-group randomized controlled trial (RCT), 16 adolescents were followed over 6 months. Data were collected at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the Cleveland metro area
* Ages 14-17 years old
* Reports moderate depressive symptoms
* Able to read, speak, and understand the English language

Exclusion Criteria:

* Current suicide risk
* Diagnosis with bipolar disorder, schizophrenia, or a personality disorder
* Severe behavioral problems that preclude group participation (as reported by parent)
* Family plans to move from the region within 6 months

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared for further analysis after main results are published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited in the community using flyers in Cleveland, Ohio from 2018-2020.
Pre-assignment Details: All consented participants were assigned arms.
Period: Overall Study
Arm/Group | Depression Management | Trust-building Self-management Together
Started | 8 | 8
3 Months Post Baseline | 8 | 8
6 Months Post Baseline | 5 | 7
Completed | 5 | 7
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed the baseline questionnaire
Groups:
- Total: Total of all reporting groups
Arm/Group | Depression Management | Trust-building Self-management Together | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.75 (0.31) | 15.13 (0.35) | 14.94 (0.23)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 1 | 6
  Transgender; Other, not specified | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 1 | 3 | 4
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) Adolescent has 8 items scored on a 4 point Likert scale summed for a total score ranging from 0-24. Higher scores indicate greater levels of depressive symptoms with a score of 10-14 indicating a moderate level of depressive symptoms. The population mean = 5.6 (SD = 1.0).
  units on a scale | 13.75 (4.03) | 12.63 (2.07) | 13.19 (3.15)
Quality of Life [Mean (Standard Deviation); unit: T-score] — The Youth Quality of Life Instrument-Short Form has 15 items measured on a 10 point Likert scale that are summed and t-scored, with higher scores indicating greater quality of life. This is a continuously distributed scale without clinical cutoff scores. The quality of life mean t-score in the population of youth without depression (M= 81.0, SD= 11.7) is greater than the mean t-score in the population of youth diagnosed with depression (M= 58.6, SD= 14.2).
  T-score | 54.75 (11.70) | 58.33 (13.59) | 56.54 (12.39)
Sleep [Mean (Standard Deviation); unit: units on a scale] — The Adolescent Sleep Hygiene Scale-revised has 8 subscales with 24 items scored on a 6 point Likert scale. Each subscale total is the mean of the items contained within. The mean of the subscale scores indicates the overall sleep score, with higher scores indicating greater sleep hygiene. The range is 1-6, with poor sleep hygiene indicated by the lowest quintile scores, which is ≤ 3.8 and good sleep hygiene is indicated by the highest quintile score, which is ≥ 4.9.
  units on a scale | 4.22 (0.85) | 4.19 (0.52) | 4.20 (0.67)
Stress management [Mean (Standard Deviation); unit: units on a scale] — The Adolescent Lifestyle Questionnaire Stress Management Subscale has four items on a 5 point Likert scale that are summed for a total score. The range is 5-20. Higher scores indicate greater stress management behavior. This is a continuously distributed scale without clinical cutoff scores. The population mean = 13.0 (SD = 3.6).
  units on a scale | 11.00 (4.28) | 10.50 (2.93) | 10.73 (3.49)
Medication adherence [Mean (Standard Deviation); unit: units on a scale] — The Extent of Non-Adherence Scale has 3 items measured on a 5-point Likert scale. A total score reflecting non-adherence is calculated by the mean of item responses. This is a continuously distributed scale without clinical cutoff scores and the range is 1-5. Greater scores indicate greater levels of non-adherence. The population mean = 1.8 (SD = 1.0).
  units on a scale | 2.08 (1.20) | 2.66 (0.33) | 2.33 (0.92)
Appointment keeping [Mean (Standard Deviation); unit: units on a scale] — The Hill-Bone Compliance Appointment Keeping Scale has 3 items measured on a four-point Likert scale. One item is reverse scored and then the three items are summed, resulting in a score ranging from 3-12. This is a continuously distributed scale without clinical cutoff scores.
  Lower scores indicate greater appointment keeping (M = 5.27 ± 0.93).
  units on a scale | 5.40 (1.81) | 6.20 (2.95) | 5.80 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-8 Adolescent
Description: The Patient Health Questionnaire-8 (PHQ-8) Adolescent has 8 items scored on a 4 point Likert scale summed for a total score ranging from 0-24. Higher scores indicate greater levels of depressive symptoms with a score of 10 indicating a moderate level of depressive symptoms. The population mean = 5.6 (SD = 1.0).
Time Frame: 3 months and 6 months post baseline
Population: Using intent-to-treat principles, all participants were included in the analysis. However, four participants were lost to follow up at 6 months post baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Depression Management: 8 weekly group sessions with self-management content
- Trust-building Self-management Together: 8 weekly group sessions with self-management content and parent relationship building content
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 6.17 (1.33) | 9.43 (6.32)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 6.80 (1.92) | 8.29 (6.40)

2. Secondary Outcome: Youth Quality of Life Scale
Description: The Youth Quality of Life Instrument-Short Form has 15 items measured on a 10 point Likert scale that are summed and t-scored, with higher scores indicating greater QoL. This is a continuously distributed scale without clinical cutoff scores. The quality of life mean t-score in the youth without depression (M= 81.0, SD= 11.7) is greater than the mean t-score in youth diagnosed with depression (M= 58.6, SD= 14.2).
Time Frame: 3 and 6 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 71.89 (18.32) | 57.33 (16.17)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 64.93 (17.10) | 61.71 (13.47)

3. Secondary Outcome: Adolescent Sleep Hygiene Scale
Description: The Adolescent Sleep Hygiene Scale-revised has 8 subscales with 24 items scored on a 6 point Likert scale. Each subscale total is the mean of the items contained within. The mean of the subscale scores indicates the overall sleep score, with higher scores indicating greater sleep hygiene. The range is 1-6, with poor sleep hygiene indicated by the lowest quintile scores, which is ≤ 3.8 and good sleep hygiene is indicated by the highest quintile score, which is ≥ 4.9.
Time Frame: 3 and 6 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 4.63 (0.62) | 4.56 (0.31)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 4.73 (0.47) | 4.17 (0.34)

4. Secondary Outcome: Stress Management
Description: The Adolescent Lifestyle Questionnaire Stress Management Subscale has four items on a 5 point Likert scale that are summed for a total score. The range is 5-20. Higher scores indicate greater stress management behavior. This is a continuously distributed scale without clinical cutoff scores. The population mean = 13.0 (SD = 3.6).
Time Frame: 3 and 6 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 14.33 (2.07) | 9.86 (1.57)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 13.40 (2.41) | 12.43 (2.15)

5. Secondary Outcome: Medication Adherence
Description: The Extent of Non-Adherence Scale has 3 items measured on a 5-point Likert scale. A total score reflecting non-adherence is calculated by the mean of item responses, with a range of 1-5. Higher scores indicate greater levels of non-adherence and lower scores indicate greater adherence. The population mean = 1.8 (SD = 1.0).
Time Frame: 3 and 6 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 2.33 (1.76) | 4.67 (0.58)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 2.08 (1.26) | 4.00 (1.41)

6. Secondary Outcome: Appointment Keeping
Description: The Hill-Bone Compliance Appointment Keeping Scale has 3 items measured on a four-point Likert scale. One item is reverse scored and then the three items are summed, resulting in a score ranging from 3-12. This is a continuously distributed scale without clinical cutoff scores. Lower scores indicate greater appointment keeping (M = 5.27 ± 0.93).
Time Frame: 3 and 6 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression Management | Trust-building Self-management Together
Number analyzed (Participants) | 8 | 8
units on a scale
  3 months post baseline | 7.40 (1.95) | 8.67 (1.53)
  6 months post baseline: number analyzed (Participants) | 5 | 7
  6 months post baseline | 7.20 (3.27) | 5.83 (2.86)

ADVERSE EVENTS:
Time Frame: Entire course of study (Baseline, 3 months, 6 months)
Arm/Group | Depression Management | Trust-building Self-management Together
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
This is a small feasibility study; therefore, these results may not be generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03599141/Prot_SAP_000.pdf